CLINICAL TRIAL: NCT04174508
Title: Evaluation of the Incidence of Diabetes Revealed at Pediatric Age in Reunion
Brief Title: Non-insulino-dependant Diabetes in Infants and Teenagers
Acronym: DIABIRUN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/CHU/10
Record Dates: First submitted 2019-11-05; First posted 2019-11-22 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Diabetes; Pediatric Disorder
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of diabetes in children, which is constantly increasing worldwide is estimated in mainland France at about 15/100 000 per year with a wide disparity between countries and a north gradient South.

In Reunion island, about 30 children a year seem to reveal diabetes before the age of 18 years but no precise data has ever been published on this subject.

Indeed, while type 1 diabetes (insulin-dependent autoimmune) represents historically the majority of cases of diabetes revealed at pediatric age (about 90%), since a little more than 10 years other types of diabetes seem emerge at pediatric age. This is particularly the case of type 2 diabetes in connection with the global epidemic of obesity.

The purpose of the investigator's study is the exhaustive prospective collection of all cases of diabetes revealed before the age of 18 in the Reunion region over a period of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* child or adolescent residing in the territory of the reunion island
* with a diagnosis that revealed diabetes according to criteria defined by WHO (World Health Organization) before 18 years of age
* Parents who signed the participation consent

Exclusion Criteria:

* Patient not residing in the usual way in Reunion island

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: child or adolescent with diabetes
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-03-24 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Average annual number of new cases of diabetes according to World Health Organization (WHO) criteria | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Laure HOUDON, MD, Principal Investigator — Centre Hospitalier Universitaire de La REUNION
Locations (4):
- France (4):
  - Groupe Hospitalier Est Réunion, Saint-Benoît
  - Centre Hospitalier Universitaire Réunion, Saint-Denis
  - Centre Hospitalier Ouest Réunion, Saint-Paul
  - Centre Hospitalier Universitaire Réunion, Saint-Pierre

IPD SHARING:
Plan to Share IPD: No